CLINICAL TRIAL: NCT02628743
Title: Multicenter, Open-Label, Single-Arm Study to Evaluate Long-Term Safety, Tolerability, and Effectiveness of 10 mg/kg BID Olesoxime in Patients With Spinal Muscular Atrophy
Brief Title: A Study to Evaluate Long Term Safety, Tolerability, and Effectiveness of Olesoxime in Patients With Spinal Muscular Atrophy (SMA)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BN29854; 2015-001589-25 (EudraCT Number)
Record Dates: First submitted 2015-12-01; First posted 2015-12-11 (Estimated); Results first posted 2019-08-09 (Actual); Last update posted 2019-08-09 (Actual); Status verified 2019-07

CONDITIONS: Muscular Atrophy, Spinal
MeSH Terms: conditions — Muscular Atrophy, Spinal | interventions — olesoxime

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Olesoxime (Experimental): Participants who have consented to the dose increase will receive 10 milligrams per kilogram (mg/kg) suspension twice a day (BID) either orally or via a naso-gastric or gastrostomy tube with breakfast and dinner, preferably at the same time of the day throughout the study. If the drug administration does not coincide with one of the scheduled meals, a snack should be taken prior to drug administration. Preferably there should be at least 10 hours between the morning and evening dose. The total dose in this study will not exceed 2000 mg.
  Participants who do not consent to the dose increase will continue with the previous dosage and receive a dose of 10 mg/kg suspension once a day orally or via a naso-gastric or gastronomy tube with the main meal, preferably at the same time of the day.
  Interventions: Drug: Olesoxime

INTERVENTIONS:
Drug: Olesoxime — Participants will receive homogeneous suspension of olesoxime.

SUMMARY:
The purpose of this open-label, single arm study is to further evaluate long-term tolerability, safety and efficacy outcomes of olesoxime in participants with Spinal Muscular Atrophy (SMA) who previously participated in one of the following two clinical studies: TRO19622 CL E Q 1115-1 (open-label Phase Ib, multicenter, single- and multiple- dose study) or TRO19622 CL E Q 1275-1 (NCT01302600, Phase II/III, adaptive, parallel-group, double blind, randomized, placebo-controlled, multicenter, multinational study).

ELIGIBILITY:
Inclusion Criteria:

* Participation in the previous studies (TRO19622 CL E Q 1115-1 or TRO19622 CL E Q 1275-1)
* For women of childbearing potential: agreement to use an acceptable birth control method during the treatment period and for at least 28 days after the last dose of olesoxime

Exclusion Criteria:

* Female participants who are pregnant or lactating, or intending to become pregnant during the study
* Participants who, in the opinion of the investigator, are not suitable to participate in this open-label study
* Participants who have developed study drug hypersensitivity to olesoxime or one of the formulation excipients, including sesame oil
* Concomitant or previous participation in any investigational drug or device study within 90 days prior to screening
* Concomitant or previous participation in a survival motor neuron 2 (SMN2) targeting antisense oligonucleotide study within 6 months prior to screening
* History of human immunodeficiency virus infection, history of Hepatitis B infection within the past year, history of Hepatitis C infection which has not been adequately treated
* History of illicit drug or alcohol abuse within 12 months prior to screening, in the investigator's judgment
* Any serious medical condition or abnormality in clinical laboratory tests that, in the investigator's judgment, precludes the participant's safe participation in and completion of the study
* History or presence of an abnormal electrocardiogram (ECG) that is clinically significant in the investigator's opinion

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2016-01-20 (Actual); Primary Completion 2018-12-18 (Actual); Study Completion 2018-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (24):
- Belgium (2):
  - UZ Gent, Ghent
  - UZ Leuven Gasthuisberg, Leuven
- France (7):
  - Hopital Femme Mere Enfant; Medecine Physique et Readaptation Pediatrique - L'ESCALE, Bron
  - Hôpital Raymond Poincare; Serv. Neurologie et Réanimation pédiatriques - Centre réf. neuromusculaire, Garches
  - Hopital Jeanne De Flandre; CIC pediatrique, Lille
  - Hopital la Timone Enfants; Service de Pediatrie et Neurologie Pediatrique, Marseille
  - CHRU de Montpellier, Hopital Gui de Chauliac; Service de Neuropediatrie, Montpellier
  - Hopital Armand Trousseau; centre reference Maladies Neuro-musculaires Est parisien Neuropediatrie, Paris
  - Hopital des Enfants; Unite de Neurologie Pediatrique, Toulouse
- Germany (3):
  - Universitätsklinikum Essen; Neuropädiatrie, Essen
  - Uniklinikum Freiburg Zentrum für Kinder- und Jugendmedizin; Neuropädiatrie und Muskelerkrankungen, Freiburg im Breisgau
  - Dr. Von Haunersches Kinderspital, München
- Italy (6):
  - Ospedale Pediatrico Bambino Gesù; Dip. Neuroscienze e Salute Mentale, Rome, Lazio
  - Policlinico Agostino Gemelli; Dipartimento di Neuropsichiatria Infantile, Rome, Lazio
  - IRCCS Istituto G. Gaslini; UOC Neurologia Pediatrica e Malattie Muscolari, Genoa, Liguria
  - I.R.C.C.S. Cà Granda - Ospedale Maggiore Policlinico; Dip. di Salute Mentale, Milan, Lombardy
  - ASST GRANDE OSPEDALE METROPOLITANO NIGUARDA;NEMO (NEuroMuscular Omnicentre);Centro clinico - Fonda, Milan, Lombardy
  - Azienda Ospedaliera Universitaria Policlinico G.Martino; Dip. Neurologia e Malattie neuromuscolari, Messina, Sicily
- UMC Utrecht; Polkliniek Neuromusculaire ziekten, Utrecht, Netherlands
- Samodzielny Publiczny Centralny Szpital Kliniczny w Warszawie; Klinika Neurologii, Warsaw, Poland
- United Kingdom (4):
  - Heart of England NHS Trust, Birmingham
  - National Hospital for Neurology and Neurosurgery,; MRC Centre for Neuromuscular Diseases, London
  - Great Ormond Street Hospital, London
  - Newcastle University & The Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne

REFERENCES:
- [Derived] Vincent-Genod D, Rippert P, Coton J, Le Goff L, Barriere A, Berruyer A, Bernard M, Garde C, Gutierrez-Garcia M, Gilabert S, Gomes-Lisboade-Souza A, Daron A, Servais L, Thomann G, Vuillerot C. Scoring People With Spinal Muscular Atrophy on the Motor Function Measure Using the Microsoft Kinect. Pediatr Phys Ther. 2023 Jan 1;35(1):36-41. doi: 10.1097/PEP.0000000000000968. Epub 2022 Oct 25. PMID 36288197

RESULTS

PARTICIPANT FLOW:
Groups:
- Olesoxime: Participants received a dose of 10 mg/kg suspension once a day (QD) orally or via a naso-gastric or gastronomy tube. Participants who consented to dose increase received 10 milligrams per kilogram (mg/kg) suspension twice a day (BID) either orally or via a naso-gastric or gastrostomy tube.
Period: Overall Study
Arm/Group | Olesoxime
Started | 131
Completed | 0
Not Completed | 131
Not completed — Other | 3
Not completed — Withdrawal by Subject | 50
Not completed — Study Terminated by Sponsor | 76
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Arm/Group | Olesoxime
Number analyzed (Participants) | 131
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.7 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66
  Male | 65
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 94
  More than one race | 0
  Unknown or Not Reported | 33
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 89
  Not Stated | 29
  Unknown | 12

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events (AEs) or Serious Adverse Events (SAEs)
Time Frame: Baseline up to approximately 3 years
Population: Safety population included all patients who received at least one dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Olesoxime
Number analyzed (Participants) | 131
percentage of participants
  SAEs | 27.5
  AEs | 91.6

2. Secondary Outcome: Change From Baseline in Motor Function Measure (MFM) Dimension 1 (D1) + Dimension 2 (D2) Score
Description: The MFM scale evaluated motor function in three dimensions. D1 evaluates functions related to standing and transfer, D2 evaluates axial and proximal function in supine and sitting position on mat and chair and D3 evaluates distal motor function. The scoring of each task uses a 4-point Likert scale based on the participant's maximal abilities without assistance: 0, cannot initiate the task or maintain the starting position; 1, performs the task partially; 2, performs the task incompletely or imperfectly (with compensatory/uncontrolled movements or slowness); and 3, performs the task fully and "normally". The scores are summed to yield a total score expressed as the percentage of the maximum possible score (the one obtained with no physical impairment); the lower the total score, the more severe the impairment.
Time Frame: Baseline (Week 1), Weeks 26, 52, 78, 104 and 130
Population: Intent-to-Treat Population (ITT) includes all participants who received at least one dose of study medication and have at least one post-baseline assessment of MFM.
Measure: Mean (Standard Deviation); unit: percentage of maximum score
Arm/Group | Olesoxime
Number analyzed (Participants) | 127
percentage of maximum score
  Baseline | 30.01 (12.77)
  Week 26 | -0.06 (4.75)
  Week 52: number analyzed (Participants) | 111
  Week 52 | -0.31 (4.61)
  Week 78: number analyzed (Participants) | 112
  Week 78 | -1.26 (5.64)
  Week 104: number analyzed (Participants) | 99
  Week 104 | -3.32 (7.08)
  Week 130: number analyzed (Participants) | 64
  Week 130 | -4.87 (9.91)

3. Secondary Outcome: Change From Baseline in MFM Total Score (D1+ D2 + Dimension 3 [D3]) Score
Description: as for outcome 2
Time Frame: Baseline (Week 1), Weeks 26, 52, 78, 104 and 130
Population: ITT population includes all participants who received at least one dose of study medication and have at least one post-baseline assessment of MFM
Measure: Mean (Standard Deviation); unit: percentage of maximum score
Arm/Group | Olesoxime
Number analyzed (Participants) | 127
percentage of maximum score
  Baseline | 41.21 (12.81)
  Week 26 | 0.31 (4.35)
  Week 52: number analyzed (Participants) | 111
  Week 52 | 0.08 (4.08)
  Week 78: number analyzed (Participants) | 112
  Week 78 | -0.64 (5.28)
  Week 104: number analyzed (Participants) | 99
  Week 104 | -2.96 (7.09)
  Week 130: number analyzed (Participants) | 64
  Week 130 | -4.02 (9.48)

4. Secondary Outcome: Plasma Concentrations of Olesoxime
Description: Values are reported separately for QD and BID doses. Dose increase occurred after Week 104.
Time Frame: Pre-dose (Hour 0) at Weeks 1, 13, 26, 39, 52, 78, 104 and 130
Population: Included participants in the safety population that received at least one dose of the study drug and had measurable concentration values.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Olesoxime
Number analyzed (Participants) | 131
ng/mL
  Baseline: number analyzed (Participants) | 128
  Baseline | 129.0 (160.2)
  Week 13: number analyzed (Participants) | 128
  Week 13 | 9475.5 (3962.5)
  Week 26: number analyzed (Participants) | 119
  Week 26 | 10021.3 (4885.6)
  Week 39: number analyzed (Participants) | 117
  Week 39 | 10257.8 (4443.7)
  Week 52: number analyzed (Participants) | 112
  Week 52 | 9665.6 (4941.8)
  Week 78: number analyzed (Participants) | 107
  Week 78 | 10351.4 (5267.3)
  Week 104: number analyzed (Participants) | 100
  Week 104 | 8566.4 (5353.1)
  Dose Increase Visit (BID): number analyzed (Participants) | 19
  Dose Increase Visit (BID) | 14797.1 (5773.8)
  Week 130 (QD): number analyzed (Participants) | 46
  Week 130 (QD) | 6274.6 (6281.9)
  Week 130 (BID): number analyzed (Participants) | 20
  Week 130 (BID) | 13956.9 (9565.0)

5. Secondary Outcome: Change From Baseline in Pediatric Quality of Life Questionnaire (PedsQL) Generic Core Scale Version 4.0 Score
Description: The PedsQL Generic Core Scale includes 23 items using self-report and/or parent report (ages 5+). The instrument covers physical, emotional, social and school functioning. Scale items are linearly transformed to a 0-100 scale (0 = 100, 1 = 75, 2 = 50, 3 = 25, and 4 = 0) so that higher scores indicate better health related quality of life.
Time Frame: Baseline (Week 1), Weeks 26, 52, 78, 104 and 130
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Olesoxime
Number analyzed (Participants) | 128
score on scale
  Baseline (Total Score) | 58.69 (11.17)
  Total Score - Week 26: number analyzed (Participants) | 126
  Total Score - Week 26 | -0.80 (9.10)
  Total Score - Week 52: number analyzed (Participants) | 118
  Total Score - Week 52 | -1.33 (10.52)
  Total Score - Week 78: number analyzed (Participants) | 109
  Total Score - Week 78 | -0.72 (10.98)
  Total Score - Week 104: number analyzed (Participants) | 101
  Total Score - Week 104 | -0.35 (11.69)
  Total Score - Week 130: number analyzed (Participants) | 67
  Total Score - Week 130 | -0.11 (10.83)
  Baseline (Physical Score) | 28.49 (16.50)
  Physical Score - Week 26: number analyzed (Participants) | 126
  Physical Score - Week 26 | -1.76 (15.99)
  Physical Score - Week 52: number analyzed (Participants) | 117
  Physical Score - Week 52 | -4.48 (17.68)
  Physical Score - Week 78: number analyzed (Participants) | 109
  Physical Score - Week 78 | -3.18 (19.67)
  Physical Score - Week 104: number analyzed (Participants) | 101
  Physical Score - Week 104 | -1.42 (17.87)
  Physical Score - Week 130: number analyzed (Participants) | 67
  Physical Score - Week 130 | -3.23 (16.33)
  Baseline (Emotional Score) | 74.61 (17.34)
  Emotional Score - Week 26: number analyzed (Participants) | 126
  Emotional Score - Week 26 | -1.19 (18.62)
  Emotional Score - Week 52: number analyzed (Participants) | 118
  Emotional Score - Week 52 | 1.19 (16.27)
  Emotional Score - Week 78: number analyzed (Participants) | 108
  Emotional Score - Week 78 | -0.05 (17.23)
  Emotional Score - Week 104: number analyzed (Participants) | 101
  Emotional Score - Week 104 | -0.54 (18.37)
  Emotional Score - Week 130: number analyzed (Participants) | 67
  Emotional Score - Week 130 | 2.31 (18.47)
  Baseline (Social Score) | 72.77 (18.59)
  Social Score - Week 26: number analyzed (Participants) | 126
  Social Score - Week 26 | 1.43 (14.15)
  Social Score - Week 52: number analyzed (Participants) | 118
  Social Score - Week 52 | 0.93 (15.91)
  Social Score - Week 78: number analyzed (Participants) | 109
  Social Score - Week 78 | 2.39 (17.38)
  Social Score - Week 104: number analyzed (Participants) | 101
  Social Score - Week 104 | 2.38 (18.62)
  Social Score - Week 130: number analyzed (Participants) | 67
  Social Score - Week 130 | 4.10 (16.05)
  Baseline (School/Work Score): number analyzed (Participants) | 127
  Baseline (School/Work Score) | 77.20 (15.83)
  School/Work Score - Week 26: number analyzed (Participants) | 125
  School/Work Score - Week 26 | -1.24 (14.28)
  School/Work Score - Week 52: number analyzed (Participants) | 117
  School/Work Score - Week 52 | -1.32 (14.09)
  School/Work Score - Week 78: number analyzed (Participants) | 107
  School/Work Score - Week 78 | -0.51 (14.26)
  School/Work Score - Week 104: number analyzed (Participants) | 100
  School/Work Score - Week 104 | -1.65 (15.24)
  School/Work Score - Week 130: number analyzed (Participants) | 66
  School/Work Score - Week 130 | -2.58 (15.04)

6. Secondary Outcome: Change From Baseline in Caregiver PedsQL Generic Core Scales Version 4.0 Score
Description: The PedsQL Generic Core Scale includes 23 items. The instrument covers physical, emotional, social and school functioning. Scale items are linearly transformed to a 0-100 scale (0 = 100, 1 = 75, 2 = 50, 3 = 25, and 4 = 0) so that higher scores indicate better health related quality of life. Questionnaire was completed by the caregiver.
Time Frame: Baseline (Week 1), Weeks 26, 52, 78, 104 and 130
Population: Intent-to-Treat Population (ITT) includes all participants who received at least one dose of study medication and have at least one post-baseline assessment of MFM. Scale scores were not computed if more than 50% of items in the scale were missing.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Olesoxime
Number analyzed (Participants) | 121
score on scale
  Baseline (Total Score) | 55.58 (12.49)
  Total Score - Week 26: number analyzed (Participants) | 115
  Total Score - Week 26 | -0.85 (13.15)
  Total Score - Week 52: number analyzed (Participants) | 106
  Total Score - Week 52 | -1.86 (13.12)
  Total Score - Week 78: number analyzed (Participants) | 103
  Total Score - Week 78 | -0.67 (13.88)
  Total Score - Week 104: number analyzed (Participants) | 93
  Total Score - Week 104 | -1.64 (17.95)
  Total Score - Week 130: number analyzed (Participants) | 62
  Total Score - Week 130 | -0.33 (13.41)
  Baseline (Physical Score) | 28.99 (25.84)
  Physical Score - Week 26: number analyzed (Participants) | 115
  Physical Score - Week 26 | -0.58 (28.66)
  Physical Score - Week 52: number analyzed (Participants) | 106
  Physical Score - Week 52 | -5.10 (25.86)
  Physical Score - Week 78: number analyzed (Participants) | 103
  Physical Score - Week 78 | -2.91 (28.91)
  Physical Score - Week 104: number analyzed (Participants) | 93
  Physical Score - Week 104 | -3.28 (34.80)
  Physical Score - Week 130: number analyzed (Participants) | 62
  Physical Score - Week 130 | -0.56 (30.09)
  Baseline (Emotional Score) | 67.48 (17.31)
  Emotional Score - Week 26: number analyzed (Participants) | 115
  Emotional Score - Week 26 | -2.13 (15.30)
  Emotional Score - Week 52: number analyzed (Participants) | 106
  Emotional Score - Week 52 | -0.90 (15.08)
  Emotional Score - Week 78: number analyzed (Participants) | 103
  Emotional Score - Week 78 | -0.39 (18.81)
  Emotional Score - Week 104: number analyzed (Participants) | 93
  Emotional Score - Week 104 | -0.70 (20.54)
  Emotional Score - Week 130: number analyzed (Participants) | 62
  Emotional Score - Week 130 | -0.32 (15.94)
  Baseline (Social Score) | 68.34 (16.19)
  Social Score - Week 26: number analyzed (Participants) | 115
  Social Score - Week 26 | -0.42 (16.84)
  Social Score - Week 52: number analyzed (Participants) | 106
  Social Score - Week 52 | -0.49 (15.92)
  Social Score - Week 78: number analyzed (Participants) | 103
  Social Score - Week 78 | 1.47 (18.40)
  Social Score - Week 104: number analyzed (Participants) | 93
  Social Score - Week 104 | -0.55 (21.72)
  Social Score - Week 130: number analyzed (Participants) | 61
  Social Score - Week 130 | 1.25 (16.22)
  Baseline (School/Work Score): number analyzed (Participants) | 120
  Baseline (School/Work Score) | 73.67 (17.69)
  School/Work Score - Week 26: number analyzed (Participants) | 112
  School/Work Score - Week 26 | -0.31 (16.69)
  School/Work Score - Week 52: number analyzed (Participants) | 104
  School/Work Score - Week 52 | 0.53 (18.14)
  School/Work Score - Week 78: number analyzed (Participants) | 101
  School/Work Score - Week 78 | 0.94 (18.39)
  School/Work Score - Week 104: number analyzed (Participants) | 91
  School/Work Score - Week 104 | -0.71 (20.64)
  School/Work Score - Week 130: number analyzed (Participants) | 59
  School/Work Score - Week 130 | -1.53 (16.17)

7. Secondary Outcome: Change From Baseline in PedsQL Neuromuscular Module Version 3.0 Scale Score
Description: The PedsQL Neuromuscular Module (Version 3.0) includes 25 items using self-report (ages 5 - 18) and/or parent report (ages 5 -18). The instrument covers problems related to neuromuscular disease, communication and family resources. Scale items are linearly transformed to a 0-100 scale (0 = 100, 1 = 75, 2 = 50, 3 = 25, and 4 = 0) so that higher scores indicate better health related quality of life.
Time Frame: Baseline (Week 1), Weeks 26, 52, 78, 104 and 130
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Olesoxime
Number analyzed (Participants) | 90
score on scale
  Baseline (Total Score) | 69.57 (14.01)
  Total Score - Week 26: number analyzed (Participants) | 89
  Total Score - Week 26 | -0.98 (10.75)
  Total Score - Week 52: number analyzed (Participants) | 81
  Total Score - Week 52 | -0.86 (12.81)
  Total Score - Week 78: number analyzed (Participants) | 79
  Total Score - Week 78 | -1.08 (12.11)
  Total Score - Week 104: number analyzed (Participants) | 70
  Total Score - Week 104 | -1.18 (13.13)
  Total Score - Week 130: number analyzed (Participants) | 52
  Total Score - Week 130 | -1.41 (12.61)
  Baseline (Neuromuscular) | 66.03 (15.39)
  Neuromuscular - Week 26: number analyzed (Participants) | 89
  Neuromuscular - Week 26 | -1.77 (12.28)
  Neuromuscular - Week 52: number analyzed (Participants) | 81
  Neuromuscular - Week 52 | -2.22 (14.29)
  Neuromuscular - Week 78: number analyzed (Participants) | 79
  Neuromuscular - Week 78 | -2.69 (12.82)
  Neuromuscular - Week 104: number analyzed (Participants) | 70
  Neuromuscular - Week 104 | -1.90 (15.11)
  Neuromuscular - Week 130: number analyzed (Participants) | 52
  Neuromuscular - Week 130 | -3.14 (14.20)
  Baseline (Family Resources Score) | 74.39 (20.10)
  Family Resources Score - Week 26: number analyzed (Participants) | 89
  Family Resources Score - Week 26 | -0.11 (17.35)
  Family Resources Score - Week 52: number analyzed (Participants) | 80
  Family Resources Score - Week 52 | 1.78 (16.07)
  Family Resources Score - Week 78: number analyzed (Participants) | 79
  Family Resources Score - Week 78 | 0.82 (19.22)
  Family Resources Score - Week 104: number analyzed (Participants) | 70
  Family Resources Score - Week 104 | -1.29 (19.81)
  Family Resources Score - Week 130: number analyzed (Participants) | 52
  Family Resources Score - Week 130 | -0.38 (16.36)
  Baseline (Communication Score) | 81.57 (21.14)
  Communication Score - Week 26: number analyzed (Participants) | 89
  Communication Score - Week 26 | 2.01 (19.86)
  Communication Score - Week 52: number analyzed (Participants) | 81
  Communication Score - Week 52 | 1.44 (24.43)
  Communication Score - Week 78: number analyzed (Participants) | 79
  Communication Score - Week 78 | 4.85 (22.19)
  Communication Score - Week 104: number analyzed (Participants) | 70
  Communication Score - Week 104 | 2.98 (24.25)
  Communication Score - Week 130: number analyzed (Participants) | 52
  Communication Score - Week 130 | 6.57 (25.15)

8. Secondary Outcome: Change From Baseline in Caregiver PedsQL Neuromuscular Module Version 3.0 Scale Score
Description: The PedsQL Neuromuscular Module (Version 3.0) includes 25 items using self-report (ages 5 - 18) and/or parent report (ages 5 -18). The instrument covers problems related to neuromuscular disease, communication and family resources. Scale items are linearly transformed to a 0-100 scale (0 = 100, 1 = 75, 2 = 50, 3 = 25, and 4 = 0) so that higher scores indicate better health related quality of life. Questionnaire was completed by the caregiver.
Time Frame: Baseline (Week 1), Weeks 26, 52, 78, 104 and 130
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Olesoxime
Number analyzed (Participants) | 88
score on scale
  Baseline (Total Score) | 59.44 (14.83)
  Total Score - Week 26: number analyzed (Participants) | 87
  Total Score - Week 26 | 0.13 (10.12)
  Total Score - Week 52: number analyzed (Participants) | 78
  Total Score - Week 52 | -0.11 (12.89)
  Total Score - Week 78: number analyzed (Participants) | 77
  Total Score - Week 78 | 0.65 (13.23)
  Total Score - Week 104: number analyzed (Participants) | 67
  Total Score - Week 104 | 1.21 (14.40)
  Total Score - Week 130: number analyzed (Participants) | 51
  Total Score - Week 130 | -0.07 (12.86)
  Baseline (Neuromuscular) | 56.28 (15.70)
  Neuromuscular - Week 26: number analyzed (Participants) | 87
  Neuromuscular - Week 26 | -0.64 (10.92)
  Neuromuscular - Week 52: number analyzed (Participants) | 78
  Neuromuscular - Week 52 | -1.33 (13.39)
  Neuromuscular - Week 78: number analyzed (Participants) | 77
  Neuromuscular - Week 78 | 0.05 (13.97)
  Neuromuscular - Week 104: number analyzed (Participants) | 67
  Neuromuscular - Week 104 | 0.54 (15.32)
  Neuromuscular - Week 130: number analyzed (Participants) | 51
  Neuromuscular - Week 130 | -1.39 (14.65)
  Baseline (Family Resources Score) | 58.24 (25.08)
  Family Resources Score - Week 26: number analyzed (Participants) | 86
  Family Resources Score - Week 26 | 1.74 (16.57)
  Family Resources Score - Week 52: number analyzed (Participants) | 77
  Family Resources Score - Week 52 | 2.44 (19.04)
  Family Resources Score - Week 78: number analyzed (Participants) | 77
  Family Resources Score - Week 78 | 0.91 (19.31)
  Family Resources Score - Week 104: number analyzed (Participants) | 67
  Family Resources Score - Week 104 | 1.27 (18.63)
  Family Resources Score - Week 130: number analyzed (Participants) | 50
  Family Resources Score - Week 130 | 1.00 (17.26)
  Baseline (Communication Score) | 79.36 (22.92)
  Communication Score - Week 26: number analyzed (Participants) | 87
  Communication Score - Week 26 | 1.92 (20.08)
  Communication Score - Week 52: number analyzed (Participants) | 78
  Communication Score - Week 52 | 2.88 (22.31)
  Communication Score - Week 78: number analyzed (Participants) | 77
  Communication Score - Week 78 | 3.57 (20.92)
  Communication Score - Week 104: number analyzed (Participants) | 67
  Communication Score - Week 104 | 4.85 (24.24)
  Communication Score - Week 130: number analyzed (Participants) | 51
  Communication Score - Week 130 | 4.90 (22.74)

9. Secondary Outcome: Change From Baseline in EuroQol 5-Dimension 5-Level (EQ-5D-5L) Questionnaire Index Score - Total Score
Description: The EQ-5D-5L is a self-reported health status questionnaire that consists of six questions used to calculate a health utility score for use in health economic analysis. There are two components to the EQ-5D-5L: a five-item health state profile that assesses mobility, self-care, usual activities, pain/discomfort, and anxiety/depression used to obtain an Index Utility Score, as well as a visual analogue scale (VAS) that measures health state. Overall scores range from 0 to 1, with low scores representing a higher level of dysfunction.
Time Frame: Baseline (Week 1), Weeks 26, 52, 78, 104 and 130
Population: Intent-to-Treat Population (ITT) includes all participants who received at least one dose of study medication and have at least one post-baseline assessment of MFM. The number analyzed represents participants who completed the questionnaire.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Olesoxime
Number analyzed (Participants) | 74
score on scale
  Baseline | 0.0471 (0.1345)
  Week 26: number analyzed (Participants) | 72
  Week 26 | 0.0084 (0.1563)
  Week 52: number analyzed (Participants) | 68
  Week 52 | -0.0164 (0.1191)
  Week 78: number analyzed (Participants) | 66
  Week 78 | 0.0168 (0.1910)
  Week 104: number analyzed (Participants) | 57
  Week 104 | 0.0081 (0.1701)
  Week 130: number analyzed (Participants) | 34
  Week 130 | -0.0259 (0.1232)

10. Secondary Outcome: Change From Baseline in Caregiver Proxy EQ-5D-5L Questionnaire Index Score - Total Score
Description: The EQ-5D-5L is a self-reported health status questionnaire that consists of six questions used to calculate a health utility score for use in health economic analysis. There are two components to the EQ-5D-5L: a five-item health state profile that assesses mobility, self-care, usual activities, pain/discomfort, and anxiety/depression used to obtain an Index Utility Score, as well as a visual analogue scale (VAS) that measures health state. Overall scores range from 0 to 1, with low scores representing a higher level of dysfunction. The questionnaire was completed by the caregiver.
Time Frame: Baseline (Week 1), Weeks 26, 52, 78, 104 and 130
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Olesoxime
Number analyzed (Participants) | 54
score on scale
  Baseline | 0.0429 (0.2335)
  Week 26: number analyzed (Participants) | 50
  Week 26 | 0.0652 (0.4091)
  Week 52: number analyzed (Participants) | 47
  Week 52 | 0.0203 (0.2820)
  Week 78: number analyzed (Participants) | 47
  Week 78 | 0.0696 (0.3094)
  Week 104: number analyzed (Participants) | 39
  Week 104 | 0.0699 (0.2887)
  Week 130: number analyzed (Participants) | 31
  Week 130 | 0.0455 (0.3323)

11. Secondary Outcome: Change From Baseline in EQ-5D-5L Visual Analogue Scale (EQ-5D-5L VAS) Score
Description: The EQ-5D-5L is a self-reported health status questionnaire that consists of six questions used to calculate a health utility score for use in health economic analysis. There are two components to the EQ-5D-5L: a five-item health state profile that assesses mobility, self-care, usual activities, pain/discomfort, and anxiety/depression used to obtain an Index Utility Score, as well as a visual analogue scale (VAS) that measures health state. The VAS is designed to rate the participant's current health state on a scale from 0 to 100, where 0 represents the worst imaginable health state and 100 represents the best imaginable health state.
Time Frame: Baseline (Week 1), Weeks 26, 52, 78, 104 and 130
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Olesoxime
Number analyzed (Participants) | 75
score on scale
  Baseline | 69.4 (19.7)
  Week 26: number analyzed (Participants) | 73
  Week 26 | 1.3 (17.1)
  Week 52: number analyzed (Participants) | 69
  Week 52 | 0.2 (17.4)
  Week 78: number analyzed (Participants) | 67
  Week 78 | 1.3 (19.9)
  Week 104: number analyzed (Participants) | 58
  Week 104 | 5.4 (17.0)
  Week 130: number analyzed (Participants) | 35
  Week 130 | 0.6 (18.1)

12. Secondary Outcome: Change From Baseline in Caregiver Proxy EQ-5D-5L VAS Score
Description: The EQ-5D-5L is a self-reported health status questionnaire that consists of six questions used to calculate a health utility score for use in health economic analysis. There are two components to the EQ-5D-5L: a five-item health state profile that assesses mobility, self-care, usual activities, pain/discomfort, and anxiety/depression used to obtain an Index Utility Score, as well as a visual analogue scale (VAS) that measures health state. The VAS is designed to rate the participant's current health state on a scale from 0 to 100, where 0 represents the worst imaginable health state and 100 represents the best imaginable health state. Questionnaire was completed by the caregiver.
Time Frame: Baseline (Week 1), Weeks 26, 52, 78, 104 and 130
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Olesoxime
Number analyzed (Participants) | 54
score on scale
  Baseline | 72.7 (21.4)
  Week 26: number analyzed (Participants) | 49
  Week 26 | -0.3 (27.7)
  Week 52: number analyzed (Participants) | 47
  Week 52 | 0.8 (21.2)
  Week 78: number analyzed (Participants) | 47
  Week 78 | 0.4 (20.9)
  Week 104: number analyzed (Participants) | 40
  Week 104 | 5.7 (24.3)
  Week 130: number analyzed (Participants) | 31
  Week 130 | 0.5 (17.9)

13. Secondary Outcome: Number of Subjects Employed Assessed Using the Work Productivity and Activity Impairment Questionnaire: Caregiver (WPAI:CG) Questionnaire
Description: The WPAI:CG consists of four questions about the effects of Spinal Muscular Atrophy (SMA) on the following: employment status, hours missed due to patient caregiving, hours missed due to other reasons, hours actually worked and two questions that measure the degree to which patient caregiving affected productivity and regular daily activities.
Time Frame: Baseline (Week 1), Weeks 26, 52, 78, 104 and 130
Population: as for outcome 9
Measure: Number; unit: participants
Arm/Group | Olesoxime
Number analyzed (Participants) | 125
participants
  Baseline: number analyzed (Participants) | 121
  Baseline | 56
  Week 26: number analyzed (Participants) | 119
  Week 26 | 66
  Week 52: number analyzed (Participants) | 109
  Week 52 | 58
  Week 78: number analyzed (Participants) | 107
  Week 78 | 62
  Week 104: number analyzed (Participants) | 97
  Week 104 | 56
  Week 130: number analyzed (Participants) | 65
  Week 130 | 39

14. Secondary Outcome: Change From Baseline in Hours Actually Worked and Work Hours Missed Assessed Using WPAI:CG Questionnaire
Description: The WPAI:CG consists of four questions about the effects of SMA on the following: employment status, hours missed due to patient caregiving (HMC), hours missed due to other reasons (HMO), hours actually worked (HAW) and two questions that measure the degree to which patient caregiving affected productivity and regular daily activities.
Time Frame: Baseline (Week 1), Weeks 26, 52, 78, 104 and 130
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Olesoxime
Number analyzed (Participants) | 56
hours
  Baseline (HMC) | 2.0 (3.7)
  HMC, Week 26: number analyzed (Participants) | 50
  HMC, Week 26 | 2.0 (7.3)
  HMC, Week 52: number analyzed (Participants) | 44
  HMC, Week 52 | 1.9 (8.2)
  HMC, Week 78: number analyzed (Participants) | 49
  HMC, Week 78 | 0.9 (5.6)
  HMC, Week 104: number analyzed (Participants) | 45
  HMC, Week 104 | 3.2 (8.3)
  HMC, Week 130: number analyzed (Participants) | 35
  HMC, Week 130 | 1.1 (8.1)
  Baseline (HMO) | 4.8 (7.3)
  HMO, Week 26: number analyzed (Participants) | 51
  HMO, Week 26 | -1.5 (7.9)
  HMO, Week 52: number analyzed (Participants) | 43
  HMO, Week 52 | -1.5 (9.0)
  HMO, Week 78: number analyzed (Participants) | 49
  HMO, Week 78 | -0.1 (8.6)
  HMO, Week 104: number analyzed (Participants) | 45
  HMO, Week 104 | 0.0 (9.6)
  HMO, Week 130: number analyzed (Participants) | 35
  HMO, Week 130 | 0.8 (7.8)
  Baseline (HAW) | 36.0 (47.0)
  HAW, Week 26: number analyzed (Participants) | 51
  HAW, Week 26 | -12.0 (46.7)
  HAW, Week 52: number analyzed (Participants) | 43
  HAW, Week 52 | -8.3 (49.2)
  HAW, Week 78: number analyzed (Participants) | 48
  HAW, Week 78 | -8.6 (49.8)
  HAW, Week 104: number analyzed (Participants) | 44
  HAW, Week 104 | 1.2 (14.4)
  HAW, Week 130: number analyzed (Participants) | 35
  HAW, Week 130 | 1.5 (27.5)

15. Secondary Outcome: Change From Baseline in Work Time Missed, Impairment While Working, Overall Work Impairment and Activity Impairment Assessed Using WPAI:CG Questionnaire Score
Description: The WPAI:CG consists of four questions about the effects of Spinal Muscular Atrophy (SMA) on the following: employment status, hours missed due to patient caregiving, hours missed due to other reasons, hours actually worked and two questions that measure the degree to which patient caregiving affected productivity and regular daily activities. WPAI:CG outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity. The outcomes are presented for Percent work time missed (WTM), Percent impairment (IMP), Percent overall work impairment (OWI) and Percent activity impairment (AIM).
Time Frame: Baseline (Week 1), Weeks 26, 52, 78, 104 and 130
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Olesoxime
Number analyzed (Participants) | 121
percentage
  Baseline (WTM): number analyzed (Participants) | 53
  Baseline (WTM) | 6.7 (11.9)
  WTM, Week 26: number analyzed (Participants) | 44
  WTM, Week 26 | 7.0 (22.3)
  WTM, Week 52: number analyzed (Participants) | 38
  WTM, Week 52 | 0.8 (15.4)
  WTM, Week 78: number analyzed (Participants) | 43
  WTM, Week 78 | 6.2 (23.3)
  WTM, Week 104: number analyzed (Participants) | 39
  WTM, Week 104 | 6.7 (20.1)
  WTM, Week 130: number analyzed (Participants) | 31
  WTM, Week 130 | 4.7 (24.4)
  Baseline (IMP): number analyzed (Participants) | 56
  Baseline (IMP) | 29.3 (26.6)
  IMP, Week 26: number analyzed (Participants) | 50
  IMP, Week 26 | -3.0 (22.8)
  IMP, Week 52: number analyzed (Participants) | 46
  IMP, Week 52 | -1.5 (27.3)
  IMP, Week 78: number analyzed (Participants) | 49
  IMP, Week 78 | -3.5 (25.0)
  IMP, Week 104: number analyzed (Participants) | 45
  IMP, Week 104 | 0.7 (22.8)
  IMP, Week 130: number analyzed (Participants) | 35
  IMP, Week 130 | -6.9 (24.7)
  Baseline (OWI): number analyzed (Participants) | 53
  Baseline (OWI) | 33.8 (28.1)
  OWI, Week 26: number analyzed (Participants) | 43
  OWI, Week 26 | -3.6 (25.3)
  OWI, Week 52: number analyzed (Participants) | 38
  OWI, Week 52 | -3.3 (25.4)
  OWI, Week 78: number analyzed (Participants) | 43
  OWI, Week 78 | -3.0 (31.9)
  OWI, Week 104: number analyzed (Participants) | 39
  OWI, Week 104 | 3.5 (26.2)
  OWI, Week 130: number analyzed (Participants) | 31
  OWI, Week 130 | -3.4 (33.3)
  Baseline (AIM) | 45.8 (29.3)
  AIM, Week 26: number analyzed (Participants) | 114
  AIM, Week 26 | -3.9 (28.7)
  AIM, Week 52: number analyzed (Participants) | 106
  AIM, Week 52 | -1.3 (30.6)
  AIM, Week 78: number analyzed (Participants) | 105
  AIM, Week 78 | -6.3 (32.6)
  AIM, Week 104: number analyzed (Participants) | 94
  AIM, Week 104 | -7.6 (27.8)
  AIM, Week 130: number analyzed (Participants) | 64
  AIM, Week 130 | -5.5 (31.7)

16. Secondary Outcome: Change From Baseline in Degree Patient Caregiving Affected Productivity and Activities Using WPAI:CG Questionnaire
Description: The WPAI:CG consists of four questions about the effects of Spinal Muscular Atrophy (SMA) on the following: employment status, hours missed due to patient caregiving, hours missed due to other reasons, hours actually worked and two questions that measure the degree to which patient caregiving affected productivity and regular daily activities. WPAI:CG outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity.
Time Frame: Baseline (Week 1), Weeks 26, 52, 78, 104 and 130
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: percentage of impairment
Arm/Group | Olesoxime
Number analyzed (Participants) | 121
percentage of impairment
  Baseline (Productivity): number analyzed (Participants) | 56
  Baseline (Productivity) | 29.3 (26.6)
  Productivity, Week 26: number analyzed (Participants) | 50
  Productivity, Week 26 | -3.0 (22.8)
  Productivity, Week 52: number analyzed (Participants) | 46
  Productivity, Week 52 | -1.5 (27.3)
  Productivity, Week 78: number analyzed (Participants) | 49
  Productivity, Week 78 | -3.5 (25.0)
  Productivity, Week 104: number analyzed (Participants) | 45
  Productivity, Week 104 | 0.7 (22.8)
  Productivity, Week 130: number analyzed (Participants) | 35
  Productivity, Week 130 | -6.9 (24.7)
  Baseline (Activities) | 45.8 (29.3)
  Activities, Week 26: number analyzed (Participants) | 114
  Activities, Week 26 | -3.9 (28.7)
  Activities, Week 52: number analyzed (Participants) | 106
  Activities, Week 52 | -1.3 (30.6)
  Activities, Week 78: number analyzed (Participants) | 105
  Activities, Week 78 | -6.3 (32.6)
  Activities, Week 104: number analyzed (Participants) | 94
  Activities, Week 104 | -7.6 (27.8)
  Activities, Week 130: number analyzed (Participants) | 64
  Activities, Week 130 | -5.5 (31.7)

17. Secondary Outcome: Change From Baseline in Short-Form 36 (SF-36) Physical Composite Scores (PCS) and Mental Composite Scores (MCS): Caregiver
Description: The SF-36 was used to assess health-related quality of life at baseline and at on-treatment visits. The SF-36 consisted of 36 questions covering 8 domains (physical functioning, role-functioning physical, bodily pain, general health, vitality, social functioning, role-functioning emotional and mental health), with each domain scoring on a scale 0-100 (a score of 0 = maximum disability and a score of 100 = no disability). The 8 domains are further summarized to 2 distinct higher-ordered clusters: the physical and mental composite t-scores (PCS and MCS). The range for all 8 domains as well as for the composite norm-based t-scores is from 0 to 100 with 100 as best possible health status and 0 as worst health status. Reported here are the Physical Composite Scores (PCS) and Mental Composite Scores (MCS).
Time Frame: Baseline (Week 1), Weeks 26, 52, 78, 104 and 130
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Olesoxime
Number analyzed (Participants) | 101
score on scale
  Baseline (PCS): number analyzed (Participants) | 99
  Baseline (PCS) | 48.07 (10.33)
  PCS, Week 26: number analyzed (Participants) | 95
  PCS, Week 26 | -0.24 (10.95)
  PCS, Week 52: number analyzed (Participants) | 87
  PCS, Week 52 | 0.27 (9.73)
  PCS, Week 78: number analyzed (Participants) | 88
  PCS, Week 78 | -0.34 (10.87)
  PCS, Week 104: number analyzed (Participants) | 77
  PCS, Week 104 | -0.48 (10.30)
  PCS, Week 130: number analyzed (Participants) | 56
  PCS, Week 130 | 1.68 (12.94)
  Baseline (MCS) | 49.71 (10.52)
  MCS, Week 26: number analyzed (Participants) | 97
  MCS, Week 26 | -1.05 (10.22)
  MCS, Week 52: number analyzed (Participants) | 89
  MCS, Week 52 | -1.64 (10.06)
  MCS, Week 78: number analyzed (Participants) | 90
  MCS, Week 78 | -0.21 (9.30)
  MCS, Week 104: number analyzed (Participants) | 79
  MCS, Week 104 | -0.08 (7.73)
  MCS, Week 130: number analyzed (Participants) | 57
  MCS, Week 130 | -1.21 (9.98)

18. Secondary Outcome: Change From Baseline in SF-36 Domain Scores: Caregiver
Description: The SF-36 was used to assess health-related quality of life at baseline and at on-treatment visits. The SF-36 consisted of 36 questions covering 8 domains (physical functioning, role-functioning physical, bodily pain, general health, vitality, social functioning, role-functioning emotional and mental health), with each domain scoring on a scale 0-100 (a score of 0 = maximum disability and a score of 100 = no disability). The range for all 8 norm-based domains was from 0 to 100 with 100 as best possible health status and 0 as worst health status.
Time Frame: Baseline (Week 1), Weeks 26, 52, 78, 104 and 130
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Olesoxime
Number analyzed (Participants) | 101
score on scale
  Baseline (Physical): number analyzed (Participants) | 99
  Baseline (Physical) | 44.51 (15.97)
  Physical, Week 26: number analyzed (Participants) | 95
  Physical, Week 26 | 1.73 (16.36)
  Physical, Week 52: number analyzed (Participants) | 87
  Physical, Week 52 | 2.03 (14.23)
  Physical, Week 78: number analyzed (Participants) | 88
  Physical, Week 78 | 1.25 (16.16)
  Physical, Week 104: number analyzed (Participants) | 77
  Physical, Week 104 | 2.39 (16.61)
  Physical, Week 130: number analyzed (Participants) | 56
  Physical, Week 130 | 6.02 (18.87)
  Baseline (Role (Physical)) | 47.95 (8.83)
  Role (physical), Week 26: number analyzed (Participants) | 97
  Role (physical), Week 26 | -1.18 (10.29)
  Role (physical), Week 52: number analyzed (Participants) | 89
  Role (physical), Week 52 | -0.76 (9.45)
  Role (physical), Week 78: number analyzed (Participants) | 90
  Role (physical), Week 78 | -1.02 (9.82)
  Role (physical), Week 104: number analyzed (Participants) | 79
  Role (physical), Week 104 | -1.05 (8.92)
  Role (physical), Week 130: number analyzed (Participants) | 57
  Role (physical), Week 130 | -0.35 (10.75)
  Baseline (Bodily pain) | 50.94 (8.77)
  Bodily pain, Week 26: number analyzed (Participants) | 97
  Bodily pain, Week 26 | -1.82 (8.75)
  Bodily pain, Week 52: number analyzed (Participants) | 89
  Bodily pain, Week 52 | -1.83 (9.04)
  Bodily pain, Week 78: number analyzed (Participants) | 90
  Bodily pain, Week 78 | -2.14 (10.55)
  Bodily pain, Week 104: number analyzed (Participants) | 79
  Bodily pain, Week 104 | -2.40 (8.44)
  Bodily pain, Week 130: number analyzed (Participants) | 57
  Bodily pain, Week 130 | -2.96 (9.82)
  Baseline (General health) | 50.21 (10.65)
  General health, Week 26: number analyzed (Participants) | 97
  General health, Week 26 | -0.63 (10.59)
  General health, Week 52: number analyzed (Participants) | 89
  General health, Week 52 | -0.75 (9.64)
  General health, Week 78: number analyzed (Participants) | 90
  General health, Week 78 | -0.22 (10.83)
  General health, Week 104: number analyzed (Participants) | 79
  General health, Week 104 | -1.17 (11.22)
  General health, Week 130: number analyzed (Participants) | 57
  General health, Week 130 | 1.07 (11.87)
  Baseline (Vitality) | 51.28 (9.42)
  Vitality, Week 26: number analyzed (Participants) | 97
  Vitality, Week 26 | -1.04 (8.48)
  Vitality, Week 52: number analyzed (Participants) | 89
  Vitality, Week 52 | -1.23 (7.53)
  Vitality, Week 78: number analyzed (Participants) | 90
  Vitality, Week 78 | -0.03 (9.67)
  Vitality, Week 104: number analyzed (Participants) | 79
  Vitality, Week 104 | -0.07 (8.16)
  Vitality, Week 130: number analyzed (Participants) | 57
  Vitality, Week 130 | 0.37 (8.57)
  Baseline (Social) | 48.01 (9.49)
  Social, Week 26: number analyzed (Participants) | 97
  Social, Week 26 | -0.67 (10.60)
  Social, Week 52: number analyzed (Participants) | 89
  Social, Week 52 | -1.24 (11.14)
  Social, Week 78: number analyzed (Participants) | 90
  Social, Week 78 | 0.28 (10.29)
  Social, Week 104: number analyzed (Participants) | 79
  Social, Week 104 | -0.95 (9.12)
  Social, Week 130: number analyzed (Participants) | 57
  Social, Week 130 | 0.35 (10.46)
  Baseline (Role (emotional)) | 48.38 (9.58)
  Role (emotional), Week 26: number analyzed (Participants) | 97
  Role (emotional), Week 26 | -1.15 (10.59)
  Role (emotional), Week 52: number analyzed (Participants) | 89
  Role (emotional), Week 52 | -1.72 (11.38)
  Role (emotional), Week 78: number analyzed (Participants) | 90
  Role (emotional), Week 78 | -1.16 (10.58)
  Role (emotional), Week 104: number analyzed (Participants) | 79
  Role (emotional), Week 104 | -1.06 (8.03)
  Role (emotional), Week 130: number analyzed (Participants) | 57
  Role (emotional), Week 130 | -0.43 (9.87)
  Baseline (Mental health) | 48.46 (9.39)
  Mental health, Week 26: number analyzed (Participants) | 97
  Mental health, Week 26 | -0.24 (9.73)
  Mental health, Week 52: number analyzed (Participants) | 89
  Mental health, Week 52 | -0.50 (9.15)
  Mental health, Week 78: number analyzed (Participants) | 90
  Mental health, Week 78 | 0.07 (7.77)
  Mental health, Week 104: number analyzed (Participants) | 79
  Mental health, Week 104 | 1.32 (7.42)
  Mental health, Week 130: number analyzed (Participants) | 57
  Mental health, Week 130 | -0.29 (9.21)

19. Secondary Outcome: Change From Baseline in Revised Utility Index Score (SF-6D_R2): Caregiver
Description: The SF-6D focuses on seven of the eight health domains covered by the SF-36: physical functioning, role participation (combined role-physical and role-emotional), social functioning, bodily pain, mental health, and vitality. SF-6D Health Utility Index (HUI) Score = 0 (worst measured health state) to 1 (best measured health state).
Time Frame: Baseline (Week 1), Weeks 26, 52, 78, 104 and 130
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Olesoxime
Number analyzed (Participants) | 98
score on scale
  Baseline | 0.70 (0.11)
  Week 26: number analyzed (Participants) | 92
  Week 26 | -0.01 (0.12)
  Week 52: number analyzed (Participants) | 86
  Week 52 | -0.01 (0.10)
  Week 78: number analyzed (Participants) | 87
  Week 78 | -0.01 (0.12)
  Week 104: number analyzed (Participants) | 76
  Week 104 | 0.00 (0.11)
  Week 130: number analyzed (Participants) | 54
  Week 130 | 0.01 (0.13)

20. Secondary Outcome: SMA Independence Scale (SMAIS) Score: Patient
Description: The SMAIS was developed specifically for SMA in order to assess function-related independence. The SMAIS contains 29 items, assessing the amount of assistance required from another individual to perform daily activities, such as eating or transferring to/from a wheelchair. Each item is scored on a zero to four scale (with an additional option to indicate that an item is non-applicable). Item scores are summed to create the total score. The range of total score is between 0 and 116. Lower scores indicate greater dependence on another individual.
Time Frame: Week 104 and Week 130
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Olesoxime
Number analyzed (Participants) | 14
score on scale
  Week 104 | 71.7 (23.4)
  Week 130: number analyzed (Participants) | 12
  Week 130 | 74.8 (22.5)

21. Secondary Outcome: SMA Independence Scale (SMAIS) Score: Caregiver
Description: as for outcome 20
Time Frame: Week 104 and Week 130
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Olesoxime
Number analyzed (Participants) | 21
score on scale
  Week 104: number analyzed (Participants) | 20
  Week 104 | 60.1 (22.2)
  Week 130: number analyzed (Participants) | 17
  Week 130 | 58.0 (24.9)

ADVERSE EVENTS:
Time Frame: Baseline up to approximately 3 years
Description: Safety population included all patients who received at least one dose of study medication.
Arm/Group | Olesoxime
All-Cause Mortality (participants affected / at risk) | 0/131
Serious Adverse Events (participants affected / at risk) | 36/131
Other Adverse Events (participants affected / at risk) | 105/131
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olesoxime (N=131)
CONSTIPATION (Gastrointestinal disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (1)
BRONCHITIS (Infections and infestations) | 3 (5)
GASTROENTERITIS (Infections and infestations) | 2 (2)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 (3)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 1 (1)
GASTRITIS (Gastrointestinal disorders) | 1 (1)
ENCEPHALITIS (Infections and infestations) | 1 (1)
GASTROINTESTINAL INFECTION (Infections and infestations) | 1 (1)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 4 (7)
LUNG INFECTION (Infections and infestations) | 2 (2)
OSTEOMYELITIS (Infections and infestations) | 1 (1)
PNEUMONIA (Infections and infestations) | 10 (13)
PNEUMONIA VIRAL (Infections and infestations) | 1 (1)
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 1 (1)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (3)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1)
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1)
PATHOLOGICAL FRACTURE (Musculoskeletal and connective tissue disorders) | 1 (1)
OBSTRUCTIVE AIRWAYS DISORDER (Respiratory, thoracic and mediastinal disorders) | 1 (1)
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 2 (4)
TESTICULAR TORSION (Reproductive system and breast disorders) | 1 (1)
MEDICAL DEVICE REMOVAL (Surgical and medical procedures) | 1 (1)
SKIN GRAFT (Surgical and medical procedures) | 1 (1)
ACCIDENTAL OVERDOSE (Injury, poisoning and procedural complications) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 1 (1)
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 2 (2)
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 1 (1)
POSTOPERATIVE WOUND COMPLICATION (Injury, poisoning and procedural complications) | 1 (1)
PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 (1)
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 1 (1)
PROCEDURAL PNEUMOTHORAX (Injury, poisoning and procedural complications) | 1 (1)
THERMAL BURN (Injury, poisoning and procedural complications) | 1 (1)
FOOD REFUSAL (Metabolism and nutrition disorders) | 1 (1)
ANXIETY (Psychiatric disorders) | 1 (1)
DEPRESSED MOOD (Psychiatric disorders) | 1 (1)
NEPHROLITHIASIS (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olesoxime (N=131)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 8 (12)
CONSTIPATION (Gastrointestinal disorders) | 9 (13)
DIARRHOEA (Gastrointestinal disorders) | 20 (34)
NAUSEA (Gastrointestinal disorders) | 9 (13)
VOMITING (Gastrointestinal disorders) | 23 (43)
PYREXIA (General disorders) | 28 (40)
BRONCHITIS (Infections and infestations) | 15 (22)
GASTROENTERITIS (Infections and infestations) | 13 (18)
INFLUENZA (Infections and infestations) | 13 (14)
NASOPHARYNGITIS (Infections and infestations) | 30 (57)
PHARYNGITIS (Infections and infestations) | 7 (9)
RHINITIS (Infections and infestations) | 10 (15)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 36 (63)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 12 (14)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 9 (16)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 8 (8)
HEADACHE (Nervous system disorders) | 23 (44)
COUGH (Respiratory, thoracic and mediastinal disorders) | 17 (23)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 16 (29)
RASH (Skin and subcutaneous tissue disorders) | 8 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2017-11-14): https://cdn.clinicaltrials.gov/large-docs/43/NCT02628743/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-15): https://cdn.clinicaltrials.gov/large-docs/43/NCT02628743/SAP_001.pdf